CLINICAL TRIAL: NCT00895960
Title: Phase I/II Trial of Dasatinib (Sprycel) With Radiation Therapy and Concomitant and Adjuvant Temozolomide in Patients With Newly-Diagnosed Glioblastoma
Brief Title: Dasatinib Plus Radiation Therapy/Temozolomide in Newly-Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew support; Study did not progress to Phase II.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0318; NCT02661113 (obsolete NCT alias)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Glioblastoma; CNS Disease; Brain Diseases
Keywords: Brain; CNS Disease; CNS; Intracranial Supratentorial GBM; Gliosarcoma; GS; Glioblastoma; GBM; Dasatinib; Sprycel; Temozolomide; TMZ; Temodar; Radiation Therapy; Radiotherapy; RT
MeSH Terms: conditions — Glioblastoma; Central Nervous System Diseases; Brain Diseases; Gliosarcoma | interventions — Dasatinib; Radiation; Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib Plus RT + TMZ (Experimental): Dasatinib (Sprycel) with Radiotherapy (RT) and 6 weeks of concomitant Temozolomide (TMZ)
  Interventions: Drug: Dasatinib; Radiation: RT (Radiotherapy); Drug: TMZ (Temozolomide)

INTERVENTIONS:
Drug: Dasatinib — Starting dose of 150 mg/day administered by mouth daily on Days 1 to 28 of every 28 day cycle, beginning on the first day of RT.
  Other Names: BMS-354825; Sprycel
Radiation: RT (Radiotherapy) — As a part of standard of care, receive 60 Gy radiation therapy Monday-Friday for a total of 30 radiation treatments (about 6 weeks).
  Other Names: Radiation Therapy
Drug: TMZ (Temozolomide) — 75 mg/m^2 capsules daily by mouth for up to a maximum of 7 weeks beginning first day of RT until RT end followed by 4 weeks off then 150 mg/m^2 daily on Days 1-5 of each 28 day study cycle and 200 mg/m^2 daily of subsequent cycles.
  Other Names: Temodar

SUMMARY:
Phase I:

Primary Objectives:

-To define the maximum tolerated dose (MTD) of dasatinib (Sprycel) with radiotherapy (RT) and 6 weeks of concomitant temozolomide (TMZ) administered at 75 mg/m^2/day in patients with newly-diagnosed glioblastoma (GBM).

Secondary Objectives:

* To characterize the safety profile of dasatinib (Sprycel) in combination with radiotherapy (RT) and concomitant TMZ in patients with newly-diagnosed GBM.
* To characterize the safety profile of dasatinib (Sprycel) in combination with adjuvant TMZ in patients with glioblastoma after RT.

STUDY DID NOT PROGRESS TO PHASE II PORTION.

Phase II:

Primary Objectives:

-To determine the effectiveness of dasatinib (Sprycel) with radiotherapy (RT) and 6 weeks of concomitant temozolomide (TMZ) administered at 75 mg/m^2/day followed by adjuvant temozolomide with concurrent dasatinib in patients with newly-diagnosed glioblastoma (GBM) as measured by overall survival.

Secondary Objectives:

* To determine the efficacy of this treatment as measured by radiographic response (RR), progression-free survival (PFS) and time to progression (TTP).
* To characterize the safety profile of dasatinib (Sprycel) in combination with RT and concomitant TMZ in patients with newly-diagnosed GBM.
* To characterize the safety profile of dasatinib (Sprycel) in combination with adjuvant TMZ in patients with GBM after RT.

Exploratory Objectives:

-To correlate tumor genotype, tumor expression of dasatinib target proteins (e.g. Src, EphA2, c-kit and PDGFR), and PTEN levels with response to therapy with dasatinib and temozolomide.

DETAILED DESCRIPTION:
PHASE I

The Study Drugs:

Dasatinib is designed to change the function of certain genes. By changing the function of these genes, it may prevent cancer from growing and spreading. It is also designed to block or lower the activity of one or more tumor-causing proteins responsible for the uncontrolled growth of tumor cells, which may result in shrinking or stopping tumor growth.

Temozolomide is designed to kill cancer cells by damaging DNA (the genetic material of cells). The damaged DNA may cause tumor cell death.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of dasatinib based on when you joined this study. Up to 2 dose levels of dasatinib will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of dasatinib given in combination with temozolomide is found.

All the groups will take the same dose level of temozolomide for the entire study.

The amount of study drugs you receive may change if you experience side effects. If at any time you experience any intolerable side effects, tell the study doctor right away.

Study Drug Administration:

During Radiation:

As a part of standard of care, you will receive radiation therapy Monday-Friday for a total of 30 radiation treatments (about 6 weeks).

Every day while you are receiving radiation, you will take the temozolomide by mouth once a day for up to a maximum of 7 weeks.

You should swallow temozolomide whole, one right after the other, without chewing them. If you vomit while taking temozolomide, you cannot take more capsules before the next scheduled dose. They should be taken on an empty stomach (at least 1 hour before and 2 hours after eating) with 1 cup (about 8 oz.) of water.

Every day while you are receiving radiation, you will take dasatinib by mouth 1 time a day for up to a maximum of 7 weeks. You should take dasatinib without food (1 hour before or 2 hours after eating), with at least 1 cup (8 oz.) of water.

After Radiation:

After the radiation therapy ends, every day, you will continually take dasatinib by mouth 1 time a day.

You will not take temozolomide for about 4 weeks after the radiation therapy ends. After 4 weeks, you will begin taking temozolomide 1 time a day, by mouth, on Days 1-5 of each 28 day study cycle.

Study Visits:

Four (4) weeks after the end of radiation, then every 4 weeks after that, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have a neurological exam.
* You will have a performance status evaluation.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* Blood (about 1 teaspoon) will be drawn to check your blood's ability to clot normally.

Every week for the first 6 weeks, then every 4 weeks after that, you will be asked if you have experienced any side effects.

If you are taking an anti-seizure drug, every 2 weeks for the first 6 weeks and then every 4 weeks after that, blood (about 1 teaspoon) will be drawn to check the levels of anti-seizure drug in your blood.

At Week 6, then before each cycle after radiation for the first 6 cycles, you will have an ECG.

Every week for the first 6 weeks, then on Days 1 and 22 of every cycle after radiation, blood (about 3 teaspoons) will be collected for routine tests.

Four (4) weeks after the end of radiation, then every 8 weeks after that, you will have an MRI scan to check the status of the disease.

Length of Study:

You may continue taking temozolomide for up to 12 cycles. You may continue taking dasatinib for as long as you are benefitting. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

End-of-Study Visit:

After you go off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will have a physical exam.
* You will have a performance status evaluation.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* You will have a neurological exam.
* Blood (about 3 1/2 teaspoons) will be collected for routine tests and to check your blood's ability to clot normally.
* If you are taking an anti-seizure drug, blood (about 1 teaspoon) will be drawn to check the level of anti-seizure drug in your blood.

Long-Term Follow-up visit:

After the end-of-study visit, the study team/staff will contact you by telephone every 3 months to check how you are doing. Each phone call will take about 5 minutes.

This is an investigational study. Temozolomide is FDA approved and commercially available for the treatment of brain tumors. Dasatinib is FDA approved and commercially available for the treatment of some types of leukemia, but it is experimental for use in brain tumors. In addition, the combination of temozolomide and dasatinib is experimental for use in brain tumors. At this time, the combination is only being used in research.

Up to 72 participants will take part in this study. Up to 72 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed histologically proven intracranial supratentorial GBM or gliosarcoma (GS) will be eligible for this protocol. Patients will not be eligible if the original histology was a grade II or III glioma and a subsequent histological diagnosis of a GBM is made.
2. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
3. Diagnosis will have been established by biopsy or resection 14-28 days prior to registration. In order to permit healing, patients should not receive Day 1 of treatment until at least 14 days after surgery.
4. Patients must not have had prior cranial RT
5. Patients must have a plan to begin partial brain RT on the same day as the first dasatinib dose and the first dose of TMZ. Radiotherapy can be performed at either MD Anderson or outside facilities. Radiotherapy must be given by external beam to a partial brain field in daily fractions of 180 to 200 cGy, to a planned total dose to the tumor of approximately 6000 cGy. Stereotactic radiosurgery and brachytherapy will not be allowed.
6. Patients must not have received prior cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy for brain tumors.
7. Patients must be >/= 18 years old.
8. A contrast enhanced brain scan should be performed within 14 days prior to registration and on a corticosteroid dose that has been stable or decreasing for at least 5 days. If the corticosteroid dose is increased between the date of imaging and registration, then a new baseline MRI/CT is required. The same type of scan, i.e., MRI or CT, must be used throughout the period of protocol treatment for tumor measurement. The use of MRI rather than CT is preferred.
9. Patients must have a Karnofsky performance status of >/= 60.
10. Patients must have adequate bone marrow function (WBC >/= 3,000/µl, ANC >/= 1,500/mm^3, platelet count of >/= 100,000/mm^3, and hemoglobin >/= 10 gm/dl), adequate liver function (SGOT, SPGT and bilirubin </= 2 times ULN), serum Na, K+, Mg^2+, phosphate and Ca^2+ >/= Lower Limit of Normal (LLN) and adequate renal function (creatinine </= 1.5 mg/dL or creatinine clearance >/= 60 cc/min/1.73 m^2) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
11. Patients must be willing to forego other cytotoxic and non-cytotoxic drug therapy against the tumor while enrolled in the study.
12. Women of childbearing potential must have a negative beta-HCG pregnancy test documented within 14 days prior to registration. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

1. Patients must not have received prior Gliadel wafers.
2. Patients must not have received any investigational agents within 30 days prior to commencing study treatment.
3. Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
4. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients with the following invasive procedures: a) Major surgical procedure, open biopsy or significant traumatic injury < 14 days prior to Day 1 therapy b) Anticipation of need for major surgical procedures during the course of the study c) Core biopsy within 7 days prior to Day 1 therapy.
7. Patients must not be pregnant/breastfeeding and must agree to practice adequate contraception. Breastfeeding should be discontinued if the mother is treated with dasatinib.
8. Patients with clinically significant cardiovascular disease: a) History of ischemic or hemorrhagic stroke within past 6 months b) Uncontrolled hypertension, defined as blood pressure >140/90 mm Hg or systolic BP >180 mm Hg if diastolic blood pressure <90 mm Hg, on at least 2 repeated determinations on separate days within past 3 months c) Myocardial infarction, CABG or unstable angina within past 6 months d) New York Heart Association grade III or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris within past 6 months
9. ( 8. continued) e) Clinically significant peripheral vascular disease within past 6 months f) Pulmonary embolism, DVT, or other thromboembolic event within past 6 months. g) Diagnosed congenital long QT syndrome h) Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) i) Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec) j) Subjects with hypokalemia or hypomagnesemia if it cannot be corrected prior to dasatinib administration
10. Evidence of bleeding diathesis or coagulopathy or INR >1.5. History of significant bleeding disorder unrelated to cancer, including: a) Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease) b) Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies) c) Ongoing or recent (</= 3 months) significant gastrointestinal bleeding
11. Patients with known HIV are ineligible for this study.
12. Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
13. Patients must not have received prior therapy with dasatinib for any indication.
14. Inclusion of Women and Minorities: Both men and women and members of all races and ethnic groups are eligible for this trial.
15. Patients on the following medication will be excluded: a) Anticonvulsants: Patients on Enzyme Inducing Anticonvulsants (EIAED) will be excluded. If patients were previously on EIAEDs that have been discontinued, patients must have been off EIAEDs for >/= 2 weeks prior to initiation of dasatinib. It should also be noted whether patients were or were not previously receiving EIAEDs and the last date of administration of EIAEDs.
16. ( 15. continued) b) Antacids: Use of H2 blockers and proton pump inhibitors is prohibited because systemic antacids (H2 inhibitors, proton pump inhibitors) decrease dasatinib absorption. Patients who require antacids should use short acting, locally active agents (e.g., Maalox, Mylanta etc.). However, these agents should not be taken within either 2 hours before or 2 hours after the dasatinib dose. This is particularly important in patients with glioblastoma who are frequently on dexamethasone and prophylactic H2 blockers or proton pump inhibitors.
17. (15. continued) c) Anticoagulants/Anti-platelets: Patients on therapeutic (treatment) dose of anticoagulants (e.g. warfarin, low molecular-weight heparin) are not eligible. Patients are not allowed to take aspirin, clopidogrel, ticlopidine, Aggrenox. Patients on prophylactic anticoagulation may be enrolled and treated on study as long as their platelet count is monitored closely and maintained at >75,000 while they are receiving Dasatinib.
18. (15. continued) d) Ibuprofen and other NSAIDS: Ibuprofen and other non-steroidal anti-inflammatory drugs (NSAIDS) can inhibit platelet function. Patients may not take ibuprofen or other NSAIDs at study entry and must have stopped these agents >/=7 days prior to starting dasatinib to allow for an appropriate wash-out period.
19. (15. continued) e) Inducers and Inhibitors of CYP3A4: Patients required to be on any of those drugs will be excluded (with the exception of Dexamethasone, but all efforts should be made to reduce the dose of dexamethasone). Patients may discontinue drug at least 7 days prior to starting dasatinib.
20. (15. continued) f) Category I drugs that are generally accepted to have a risk of causing Torsades de Pointes including: (Patients must discontinue drug at least 7 days prior to starting dasatinib) (1). quinidine, procainamide, disopyramide (2). amiodarone, sotalol, ibutilide, dofetilide (3). erythromycin, clarithromycin (4). chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide (5). cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-05-07 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline then after each 28-day study cycle
  The MTD of dasatinib will be that dose at which fewer than one-third of participants experience dose limiting toxicity (DLT). Escalations are planned in groups of three patients, with an additional three patients to be added at the first indication of DLT.

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline till participant death or end of follow-up period, approximately 12 to 18 months (following 12 cycles of treatment)
  Overall survival (OS) is defined as the time from surgical diagnosis to the date of death from any cause. For participants who are still alive at the time of analysis, survival time will be censored at the last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: John De Groot, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org